CLINICAL TRIAL: NCT03727217
Title: Performance of Ultrasound in the Early Diagnosis of Vocal Cords Paralysis After Thyroidectomy or Parathyroidectomy (PECV)
Brief Title: Performance of Ultrasound in the Early Diagnosis of Vocal Cords Paralysis
Acronym: PECV
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lille Catholic University (Other)
Collaborators: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: RC-P0068
Record Dates: First submitted 2018-10-31; First posted 2018-11-01 (Actual); Last update posted 2021-02-03 (Actual); Status verified 2021-02

CONDITIONS: Thyroidectomy; Paralysis of Vocal Cords
Keywords: Thyroidectomy; Paralysis of Vocal Cords; Ultrasound
MeSH Terms: conditions — Vocal Cord Paralysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pre and postoperative ultrasound (Experimental): An ultrasound is performed in preoperative and in postoperative.
  Interventions: Diagnostic Test: Pre and postoperative ultrasound

INTERVENTIONS:
Diagnostic Test: Pre and postoperative ultrasound — An ultrasound is performed in preoperative and in postoperative

SUMMARY:
Thyroid and parathyroid surgery concerns around 50 000 patients a year in France. One of its main complications is paralysis of vocal cords, and the consequences can be serious.

In this study, the main gold is to evaluate diagnostic performances of ultrasound for an early diagnosis (as soon as awakening of the patient) of vocal cords paralysis in the post-operative period in order to prevent at best complications.

DETAILED DESCRIPTION:
Thyroid and parathyroid surgery concerns around 50 000 patients a year in France. One of its main complications is paralysis of vocal cords. Indeed, the anatomy of the thyroid and its close location with the recurrent laryngeal nerve (responsible for the vocal cord movement) involves a possible lesion or inflammation of the nerve during the surgical procedure. This complication is common, affecting around 10% of thyroid or parathyroid patients following surgery. This complication can be reversible, with a speech therapy or a specific endoscopic treatment by an otolaryngologist.

Currently, a postoperative screening is performed by nasofibroscopy in the recovery room to directly visualize vocal cord mobility. This examination may be painful or badly tolerated by some patients.

Recent studies have highlighted the performance of ultrasound in this diagnosis. The protocol for these studies included an ultrasound distant of the intervention, while it is known that vocal cord paralysis may have earlier consequences.

In this study, the investigators would like to evaluate diagnostic performances of vocal cords ultrasound for an early diagnosis (as soon as awakening of the patient) of vocal cords paralysis in the post-operative period in order to prevent at best complications.

The main limitation of vocal cord ultrasound is mainly related to surgery. Surgery creates anatomical rearrangements, so the secondary objective of this study will be to test whether the preoperative visualization is predictive of a good postoperative visualization.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years
* Scheduled surgery of total or partial thyroidectomy or parathyroidectomy
* Patient been informed and given his/her written consent to participate
* Patient affiliated to a social security scheme

Exclusion Criteria:

- Patient under tutorship or curatorship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 113 (Actual)
Dates: Start 2018-07-10 (Actual); Primary Completion 2020-08-24 (Actual); Study Completion 2020-08-24 (Actual)

PRIMARY OUTCOMES:
Diagnostic performance comparison between ultrasound and nasofibroscopy | one hour after surgery
  Diagnostic performances (sensitivity, specificity, positive and negative predictive value) of the immediate postoperative ultrasound (within one hour after the end of surgery), the gold standard being nasofibroscopy.

SECONDARY OUTCOMES:
Frequency distribution of quality of ultrasound visualization (good or bad) measured by contingency tables | before surgery (same day), one hour after surgery
  Link between the good visualization of the vocal cords by preoperative ultrasound and postoperative ultrasound.
Time for performing ultrasound | one hour after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Claire Texier, Dr, Principal Investigator — Lille Catholic University
Locations (1):
- Lille Catholic Hospitals, Lomme, Nord, France

IPD SHARING:
Plan to Share IPD: No